CLINICAL TRIAL: NCT04562675
Title: Long-term Effects of a Lay Health Advisor Intervention on Immigrant Children's Caries: A Randomized Controlled Trial
Brief Title: Long-term Effects of a Lay Health Advisor Intervention on Immigrant Children's Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KMUHIRB-2014-04-05(Ⅰ)
Record Dates: First submitted 2020-09-14; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Caries,Dental
Keywords: Caries; immigrant; Lay health advisor; preventive behavior; oral hygiene
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (IG) (Experimental): LHA intervention group (IG)
  Interventions: Behavioral: LHA intervention
- Control group (CG) (Placebo Comparator): brochure-only control group (CG)
  Interventions: Other: brochure-only

INTERVENTIONS:
Behavioral: LHA intervention — For the IG, a 4-hour lesson consisting of 4 chapters and leaflets was delivered over 4 weeks, with one chapter per hour per week. Each LHA visited the assigned mother in the IG four times in a 4-week period.
  Arms: Intervention group (IG)
Other: brochure-only — brochure-only for control group (CG)
  Arms: Control group (CG)

SUMMARY:
The aim of this study was to evaluate the long-term effectiveness of a lay health advisor (LHA) intervention on immigrant children's caries and preventive behaviors.This randomized controlled trial included mother-child pairs in the intervention group (IG) and a brochure-only control group (CG), respectively. The IG received a four-week one-on-one session by an LHA on caries-related knowledge and brushing techniques. Baseline and follow-up surveys were used to collect the data in caries experience and maternal caries preventive behavior.

DETAILED DESCRIPTION:
A randomized experimental design was used. Vietnamese women whose children aged 2-6 years were recruited through churches, Chinese schools, immigrant service centers, kindergarten, or recommendations from LHAs in Kaohsiung City in Taiwan. Overall, 30 and 25 Vietnamese mother-child pairs were randomized into the IG and CG. G*Power (version 3.1.9.4) was used for power analysis. A power analysis was established by effect size as the mean difference of filled teeth change between baseline and 8-month follow-up measurement between the IG and CG, with sample size and 0.05 alpha level. The power was greater than 0.802, and research results have adequate power.All children underwent oral examination at baseline and at 1-week, 2- and 8-month follow-ups. Each child was examined by a dentist in accordance with the primary dentition caries experience.Each immigrant mother completed surveys at baseline and at 1-week and 8-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Vietnamese women whose children aged 2-6 years

Exclusion Criteria:

* None

Ages: 22 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2012-08-27 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
dmft index | Change from Baseline dmft at 1 weeks after intervention
  The caries status of each tooth was recorded using the dmft index, as follows: decayed (d), missing (m), or filled (f) tooth (t). For each child, caries experience was measured using the dmft index of primary teeth.
dmft index | Change from Baseline dmft at 2 months after intervention
  The caries status of each tooth was recorded using the dmft index, as follows: decayed (d), missing (m), or filled (f) tooth (t). For each child, caries experience was measured using the dmft index of primary teeth.
dmft index | Change from Baseline dmft at 8 months after intervention
  The caries status of each tooth was recorded using the dmft index, as follows: decayed (d), missing (m), or filled (f) tooth (t). For each child, caries experience was measured using the dmft index of primary teeth.

SECONDARY OUTCOMES:
Maternal preventive behavior | Change from Baseline at 1 weeks after intervention
  Item including that"Do you ask your child to brush his/her teeth?" The response was coded as zero (not/seldom/sometimes) or one (always). "How many times you help your child to brush his/her teeth every day?" The response was coded as zero (no/less than two times/day) or one (two or more times/day). "How long do you help your child brush his/her teeth every time?" The response was coded as zero (no/less than three minutes) or one (three or more minutes). "When was the last time that you took your child for a dental visit?" and "Why did you take your child for a dental visit?" The responses were coded as zero (last dental visit more than six months or dental visit for oral or tooth discomfort) or one (last dental visit six months or less and dental visit for regular checkup).
Maternal preventive behavior | Change from Baseline at 8 months after intervention
  Item including that"Do you ask your child to brush his/her teeth?" The response was coded as zero (not/seldom/sometimes) or one (always). "How many times you help your child to brush his/her teeth every day?" The response was coded as zero (no/less than two times/day) or one (two or more times/day). "How long do you help your child brush his/her teeth every time?" The response was coded as zero (no/less than three minutes) or one (three or more minutes). "When was the last time that you took your child for a dental visit?" and "Why did you take your child for a dental visit?" The responses were coded as zero (last dental visit more than six months or dental visit for oral or tooth discomfort) or one (last dental visit six months or less and dental visit for regular checkup).
Maternal caries-related knowledge | Change from Baseline at 1 weeks after intervention
  Maternal caries preventive behaviors toward children were collected by questionnaire.Ten statements were used to evaluate mothers' caries preventive knowledge, such as "Dental plaque is a major factor for oral disease" and "The Bureau of National Health Insurance (BNHI) provides children with fluoride varnish twice a year." Possible scores ranged from zero to ten, with higher scores indicating a higher level of caries preventive knowledge. The Kuder-Richardson reliability test was 0.72 for this scale.
Maternal caries-related knowledge | Change from Baseline at 8 months after intervention
  Maternal caries preventive behaviors toward children were collected by questionnaire.Ten statements were used to evaluate mothers' caries preventive knowledge, such as "Dental plaque is a major factor for oral disease" and "The Bureau of National Health Insurance (BNHI) provides children with fluoride varnish twice a year." Possible scores ranged from zero to ten, with higher scores indicating a higher level of caries preventive knowledge. The Kuder-Richardson reliability test was 0.72 for this scale.
Maternal attitude toward oral hygiene | Change from Baseline at 1 weeks after intervention
  Maternal attitude toward oral hygiene were collect by questionnaire.Eleven statements measured mothers' attitude toward their children's oral hygiene, based on the research by Skeie et al. The responses were rated on a five-point Likert-scale ranging from one ("strongly disagree") to five ("strongly agree"), with the total possible score ranging from 11 to 55. Higher scores indicated more positive attitudes toward children's oral hygiene. Cronbach's α was 0.84 for this scale.
Maternal attitude toward oral hygiene | Change from Baseline at 8 months after intervention
  Maternal attitude toward oral hygiene were collect by questionnaire.Eleven statements measured mothers' attitude toward their children's oral hygiene, based on the research by Skeie et al. The responses were rated on a five-point Likert-scale ranging from one ("strongly disagree") to five ("strongly agree"), with the total possible score ranging from 11 to 55. Higher scores indicated more positive attitudes toward children's oral hygiene. Cronbach's α was 0.84 for this scale.
Maternal self-efficacy toward oral hygiene | Change from Baseline at 1 weeks after intervention
  The following three statements were used to evaluate mothers' self-efficacy toward children's oral hygiene, based on the research by Hsu et al. "It is easy for me to help my children brush their teeth"; "I can help my children brush their teeth before bedtime" and "I can take my children to visit a dentist regularly." The scores ranged from one ("strongly disagree") to four ("strongly agree"), with the total possible score ranging from three to twelve. High scores meant that mothers were confident that they could appropriately manage their children's oral hygiene behaviors. Cronbach's α was 0.72 for this scale.
Maternal self-efficacy toward oral hygiene | Change from Baseline at 8 months after intervention
  The following three statements were used to evaluate mothers' self-efficacy toward children's oral hygiene, based on the research by Hsu et al. "It is easy for me to help my children brush their teeth"; "I can help my children brush their teeth before bedtime" and "I can take my children to visit a dentist regularly." The scores ranged from one ("strongly disagree") to four ("strongly agree"), with the total possible score ranging from three to twelve. High scores meant that mothers were confident that they could appropriately manage their children's oral hygiene behaviors. Cronbach's α was 0.72 for this scale.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Ling Huang, Principal Investigator — Kaohsiung Medical University

IPD SHARING:
Plan to Share IPD: No